CLINICAL TRIAL: NCT00997295
Title: The Effects of a Heat and Moisture Exchanger on Temperature and Humidity in Low -Flow Anesthesia Workstation
Brief Title: Heat and Moisture Exchanger and Low-flow Gas
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Clinical Research Ethic Committee of Botucatu Medical School, Botucatu Medical School, UNESP
Other Study IDs: upeclin/HC/FMB-Unesp-29
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2009-10-19 (Estimated); Status verified 2009-10

CONDITIONS: Gynecological Surgery; General Anesthesia
Keywords: low flow gas; Heat and moisture exchanger; Humidity; Temperature; Core temperature; Women

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Heat moisture exchanger (HME): This group was submitted to general anesthesia with low flow gas and heat moisture exchanger
- Low flow gas (LFG): This group was submitted to general anesthesia with only low flow gas
- Humidity of the respiration: Heat and moisture group:
  The first group (G1)will be submitted to low flow gas anesthesia and heat and moisture exchanger (HME)
  Control group:
  The second group(G2)Will be submitted to low flow gas anesthesia
- HME and LFG

SUMMARY:
The aim of the present study was to measure the inspired gas temperature and humidity of the anesthetic circuit in the Dräger Primus machine and esophageal temperature with or without and heat and moisture exchanger (HME) and low-flow gas during anesthesia in patients submitted to gynecological surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18 to 69 years old
* Gynecological

Exclusion Criteria:

* Obesity
* Fever
* Endocrine disease

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty adult patients scheduled to gynecologic surgeries were randomly assigned in two groups to received fresh gas flow of 1 l.min-1 with or without in circle anesthesia system. Relative humidity, absolute humidity, temperature of gases and esophageal temperature were measured at 15 min (T0)after respiratory circuit installation and then every 30 min up to 120 min afterwards.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jair Castro Jr, MD, Principal Investigator — Botucatu Medical Faculty
Locations (1):
- College of Medicine of Botucatu, Botucatu, São Paulo, Brazil

REFERENCES:
- [Derived] de Castro J Jr, Bolfi F, de Carvalho LR, Braz JR. The temperature and humidity in a low-flow anesthesia workstation with and without a heat and moisture exchanger. Anesth Analg. 2011 Sep;113(3):534-8. doi: 10.1213/ANE.0b013e31822402df. Epub 2011 Jun 16. PMID 21680862